CLINICAL TRIAL: NCT00006186
Title: Autologous Fresh Whole Blood and Coagulation Following Cardiopulmonary Bypass in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCRR-M01RR00069-0621; M01RR000069 (NIH)
Record Dates: First submitted 2000-08-25; First posted 2000-08-28 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Congenital Heart Defects
Keywords: dilutional coagulopathy
MeSH Terms: conditions — Heart Defects, Congenital

INTERVENTIONS:
Procedure: Autologous fresh whole blood

SUMMARY:
Dilution of blood caused by cardiopulmonary bypass (the heart-lung machine) during open heart surgery is associated with decreased concentrations in the blood of coagulation factors. This can be extreme in infants because of their small blood volumes and can lead to impairment of the normal blood clotting mechanism and excessive bleeding after the operation. Transfusion of fresh whole blood has been shown to be an effective treatment because fresh blood is rich in coagulation factors. However, it is difficult to obtain truly fresh blood from a blood bank. We hypothesized that fresh blood drawn from the patient and given back after cardiopulmonary bypass would improve the clotting mechanism. In our study, the infants in the treatment group have some of their own fresh blood removed after they are anesthetized for the operation and before they are placed on cardiopulmonary bypass. This blood is then given back to them after completion of cardiopulmonary bypass. Infants in the control group will not have their own blood removed but will undergo cardiopulmonary bypass. We will compare the two groups by drawing blood samples that measure coagulation tests.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing non-complex open heart surgery
* Diagnosis of congenital heart disease
* No previous open heart surgery
* Weight 15 kg or less

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, Denver, Colorado, United States